CLINICAL TRIAL: NCT03416192
Title: 12 Weeks of Hemodialysis With Medium Cut-Off Filter Compared to Hemodiafiltration With Standard High-flux Filter.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Capacity shortage
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2017/830/2
Record Dates: First submitted 2018-01-23; First posted 2018-01-31 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Chronic Kidney Diseases; Uremia
Keywords: Dialysis; MCO; Middle molecules
MeSH Terms: conditions — Renal Insufficiency, Chronic; Uremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MCO-HD (Experimental): Hemodialysis with Medium Cut-Off filter
  Interventions: Device: MCO-HD; Device: high-flux HDF
- High-flux HDF (Active Comparator): Hemodiafiltration with standard high-flux filter
  Interventions: Device: MCO-HD; Device: high-flux HDF

INTERVENTIONS:
Device: MCO-HD — Measurements will be done after 0,4,8 and 12 weeks of hemodialysis with Medium Cut-Off filter.
Device: high-flux HDF — Measurements will be done after 0,4,8 and 12 weeks of hemodiafiltration with standard high-flux filter

SUMMARY:
The medium cut-off dialysis (MCO) membrane has been developed to improve middle molecule removal compared to standard high-flux dialysis filters.

The aim of this study is to compare levels of middle molecules after 12 weeks of MCO hemodialysis, compared to 12 weeks of hemodiafiltration using standard high-flux filter.

ELIGIBILITY:
Inclusion Criteria:

* Ongoing HDF treatment (>3 months)
* Oliguric
* Albumin ≥ 30
* CRP <15
* No acute myocardial infarction within 3 months.
* Swedish or english speaking.

Exclusion Criteria:

- Not able to understand the study information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of predialysis mean of middle molecules after 12 weeks (Beta-2-microglobulin, Cystatin C, Myoglobin, Beta-Trace Protein, Troponin T, Prealbumin). | 12 weeks
Comparison of postdialysis mean of middle molecules after 12 weeks (Beta-2-microglobulin, Cystatin C, Myoglobin, Beta-Trace Protein, Troponin T, Prealbumin). | 12 weeks

SECONDARY OUTCOMES:
Comparison of predialysis mean of small molecules (CRP, Urea, Phosphate and Creatinine) after 12 weeks. | 12 weeks
Comparison of postdialysis mean of of small molecules (CRP, Urea, Phosphate and Creatinine) after 12 weeks. | 12 weeks
Comparison of predialysis mean of large molecules after 12 weeks (Albumin, Transferrin, IgG). | 12 weeks
Comparison of postdialysis mean of large molecules after 12 weeks (Albumin, Transferrin, IgG). | 12 weeks
Comparison of pre- and postdialysis mean of all molecules at 0, 4 and 8 weeks. | 8 weeks
Comparison of number of adverse effects during the study period. | 12 weeks
Comparison of mean nPCR after 12 weeks. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anders Christensson, MD, PhD, Principal Investigator — Region Skane, Lund University

IPD SHARING:
Plan to Share IPD: No